CLINICAL TRIAL: NCT01753934
Title: Diabetic Ketoacidosis and Its Impact on Neurocognition
Brief Title: Diabetic Ketoacidosis and Its Impact on the Brain
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: William E And Aenid R Weisgerber Foundation (Other)
Responsible Party: Principal Investigator, Tandy Aye, Assistant Professor, Stanford University
Other Study IDs: SU-05102011-7713
Record Dates: First submitted 2012-09-18; First posted 2012-12-20 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — There is no intervention. All subjects with DM and controls get neurocognitive testing and an MRI of the brain. We want to see if the scores are different but no changes in therapy will be done.
Oversight: Data Monitoring Committee: No

SUMMARY:
About the Study: This research study is being conducted to see if diabetic ketoacidosis has any impact on learning, behavior and development in children with Type 1 diabetes mellitus. If there is an impact, is it transient or persistent? Sixty to 80 children between the ages of 4 to 17 years with Type 1 diabetes mellitus will have neuropsychological testing and a non-sedated MRI scan of the head performed. The investigators will compare this to a control group of 30-40 children between the ages of 4 to 17 years without Type 1 diabetes mellitus. The children with Type 1 diabetes mellitus will not have any changes made to their current diabetes regimen. The children with Type 1 diabetes mellitus should continue to check blood glucose values as required by your doctor and bring their meter(s) for downloading to each visit. The children with Type 1 diabetes mellitus should also tell your doctor about the frequency of severe low and high blood glucose values.

DETAILED DESCRIPTION:
Participant Schedule:

1. One visit for 3-4 hours at the Stanford Medical Center to complete neuropsychological testing and to become familiar with the MRI scanner.
2. Subjects who need to become more familiar with the MRI scanning process will view a video tape at home.
3. One visit for 1-2 hours at Stanford Medical Center to have the MRI scan of the head completed.
4. Subjects between 10 and 17 years of age will also be asked to complete two additional abbreviated neuropsychological tests at one week and one month from enrollment.
5. Subjects may have the complete neuropsychological testing and MRI scan repeated 15 months from time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

To take part in the study, the participant must meet the following inclusion criteria:

1. Be between the ages of 4 to 17 years.
2. Either has been diagnosed with type 1 diabetes mellitus OR does not have type 1 diabetes mellitus

Exclusion Criteria:

If the interested participant has a history of head trauma with any loss of consciousness, prematurity (born less than 30 weeks of gestation), significant developmental delay (lack of single word speech or ability to walk independently by 18 months of age), neurologic disease independent of diabetes (eg seizure disorder or medical contraindication to MRI procedure (eg metal appliances such as braces).

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sixty to 80 children between the ages of 4 to 17 years with Type 1 diabetes mellitus will have neuropsychological testing and a non-sedated MRI scan of the head performed. We will compare this to a control group of 30-40 children between the ages of 4 to 17 years without Type 1 diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Memory score on ImPACT testing | 15 months
  The computerized electronic testing generates a standardized test score at the complete of the test. The scores will be compared from enrollment, one week, one month and at 3 months. The change in score from enrollment to one week with be the main number used for analysis

SECONDARY OUTCOMES:
White matter volume on MRI using diffusion tensor imaging | 15 months
  Values will be calculated according to manuscript by Aye et al in Diabetes Care Sept 2012 electronically published ahead; available on line

CONTACTS AND LOCATIONS:
Overall Officials: Tandy Aye MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Aye T, Mazaika PK, Mauras N, Marzelli MJ, Shen H, Hershey T, Cato A, Weinzimer SA, White NH, Tsalikian E, Jo B, Reiss AL; Diabetes Research in Children Network (DirecNet) Study Group. Impact of Early Diabetic Ketoacidosis on the Developing Brain. Diabetes Care. 2019 Mar;42(3):443-449. doi: 10.2337/dc18-1405. Epub 2018 Dec 20. PMID 30573652